CLINICAL TRIAL: NCT06192394
Title: Effect of Gum Chewing or Walking Exercise on the Quality of Bowel Preparation and Patient Satisfaction Compared to Standard Preparation Before Colonoscopy
Brief Title: Effect of Gum Chewing or Walking on Bowel Prep Quality and Patient Satisfaction Before Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, ibrahim kiyat, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IUC-HEM-IK-01
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: Colonoscopy; Patient Satisfaction; Chewing Gum; Walking Exercise
MeSH Terms: conditions — Patient Satisfaction | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: There are three groups: control, gum chewing and walking exercise.
Who Masked: Care Provider
Masking Description: On the day of the colonoscopy procedure, endoscopy nurses and physicians (single blind) will not know which group the patients are in. Patients will be asked not to share information about which group they will be in with the endoscopy team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Sham Comparator): Patients in the control group will undergo the standard bowel preparation determined by the hospital, which includes the following steps:
  * No solid food should be consumed after the evening meal 2 days before colonoscopy.
  * Only clear liquids should be consumed the day before colonoscopy.
  * If the colonoscopy is scheduled for 12:00 PM, nothing should be eaten or drank after midnight on the preceding night; if the colonoscopy is scheduled for the afternoon, nothing should be consumed after 06:00 AM on the same day.
  * The entire X-M Diet syrup should be consumed with plenty of water within 1 hour at 4:00 PM and 8:00 PM the day before colonoscopy. Additionally, an enema (BT Enema) should be administered at 11:00 PM the night before and at 07:00 AM on the day of colonoscopy.
  Interventions: Other: Control
- Chewing Gum Group (Active Comparator): All patients in the gum-chewing group will receive the following interventions in addition to standard bowel preparation:
  * Patients will be instructed to chew xylitol gum for 20 minutes at three intervals (17:00-19:00, 19:00-21:00, 21:00-23:00) after consuming the prescribed X-M Diet syrup on the day before the procedure.
  * Following the administration of an enema on the procedure day, patients will be instructed to chew gum every 2 hours for 20 minutes until one hour before the scheduled procedure time.
  Interventions: Other: Chewing Gum
- Walking Exercise Group (Active Comparator): All patients in the walking group will receive the following interventions in addition to standard bowel preparation:
  * Patients will be asked to drink the prescribed X-M diet syrup 1 day before the procedure and then walk for 1 hour at two specific times (from 18:00 to 19:00 and from 22:00 to 23:00).
  * On the day of the procedure, after the enema, patients will be instructed to walk from 08:00 until one hour before the scheduled procedure time.
  * Patients will be given a pedometer to count their steps and will be asked to walk at least 3000 steps before the colonoscopy procedure.
  Interventions: Other: Walking Exercise

INTERVENTIONS:
Other: Chewing Gum — Patients will be asked to chew xylitol gum for 20 minutes every 2 hours (17.00-19.00, 19.00-21.00, 21.00-23.00) after drinking the X-M Diet syrup prescribed the day before the colonoscopy procedure. After the enema is given on the day of the colonoscopy, they will be asked to chew gum for 20 minutes every 2 hours until one hour before the scheduled procedure time. Xylitol is a naturally occurring five-carbon sugar alcohol (C5H12O5) found in fruits and vegetables such as plums, strawberries, cauliflower, and pumpkin. It is similar in taste to sucrose but contains 40% fewer calories than other carbohydrates (1 gram of xylitol = 2.4 calories). Xylitol has positive effects on dental health and may also have beneficial impacts on other systems such as immunity, respiratory, and digestive systems. Since xylitol is not digested by human enzymes, it has a laxative effect. In the study, sugar-free gum with xylitol will be used.
  Arms: Chewing Gum Group
Other: Walking Exercise — Patients will be given a pedometer to count their steps and will be asked to walk at least 3000 steps before the colonoscopy procedure.
  Arms: Walking Exercise Group
Other: Control — Patients will undergo standard bowel preparation determined by the hospital.
  Arms: Control Group

SUMMARY:
Colorectal cancers are a major global health problem, highlighting the critical importance of screening programs for early diagnosis and effective treatment. The success of colonoscopy largely depends on the quality of bowel preparation. Inadequate bowel preparation may reduce the effectiveness of colonoscopy and cause lesions to be missed.

Previous research has shown the positive effects of diet, training, and polyethylene glycol use on bowel readiness. However, there is limited research on the effects of methods such as gum chewing and walking exercise.

This study aims to evaluate the effects of gum chewing and walking exercise, as well as diet and medication, on the quality of bowel preparation and patient satisfaction during the bowel preparation process before colonoscopy. The study uses a randomized controlled, single-blind experimental design with three different groups: a control group, a gum chewing group, and a walking exercise group. Each group will be evaluated based on bowel preparation quality and patient satisfaction. The quality of bowel preparation will be determined using the Boston Bowel Preparation Scale, and factors such as polyp detection, workability of colonoscopy, and cecal intubation time will also be evaluated. Patient satisfaction levels will be evaluated by taking into account how satisfied the patients are with the colonoscopy procedure and their complaints before and after the procedure.

The results of this study will contribute to a better understanding of the impact of chewing gum and walking exercise before colonoscopy on the quality of bowel preparation and patient satisfaction. Identifying effective methods to improve the quality of bowel preparation can contribute to a healthier society by raising the standard of nursing care. At the same time, this research may improve the comfort and effectiveness of the colonoscopy process for patients and benefit public health by increasing the effectiveness of colorectal cancer screening programs.

DETAILED DESCRIPTION:
An ideal bowel preparation should have the capacity to evacuate the fecal load quickly, without compromising the comfort of patients or causing fluid-electrolyte imbalance. Various methods are used to improve the quality of bowel preparation, such as pre-colonoscopy education, low-fiber diet, and use of split-dose polyethylene glycol (PEG). There are many scientific studies showing that these methods increase the quality of bowel preparation. However, there have been fewer studies showing that methods such as chewing gum and walking exercises before colonoscopy increase the quality of bowel preparation. No study has been found in which these two methods were evaluated together. In order to eliminate the deficiency in this field, it is thought that this study will be useful in improving the quality of bowel preparation before colonoscopy.

Chewing gum is a virtual feeding method that stimulates the cephalic-vagal reflex, promoting the secretion of gastric and intestinal hormones and increasing intestinal motility. Chewing gum has advantages such as ease of application, low cost, and no reported side effects. Therefore, the use of this method as a safe intervention is recommended. Its effectiveness in reducing postoperative ileus and hospital stay has been demonstrated in many studies.

It is stated that walking exercise improves bowel cleanliness and reduces discomfort associated with nausea and abdominal pain during bowel preparation for colonoscopy. A systematic review found that low and moderate-intensity exercise lasting less than 60 minutes supports gastrointestinal motility.

Inadequate bowel preparation can lead to the repetition of the colonoscopy procedure, negatively affecting patients' experiences and satisfaction. In addition to this, factors such as the difficulty of the bowel preparation process in patients undergoing colonoscopy, unsedated colonoscopy, long appointment dates, and insufficient pre-procedure information can also negatively impact patient satisfaction. Assessing the satisfaction of patients is recommended for a successful and high-quality colonoscopy procedure.

This study was designed as a randomized controlled experimental study to determine the effects of gum chewing and walking exercise, as well as the use of diet and medication during the bowel preparation process before colonoscopy, on the quality of bowel preparation and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65 years,
* Capable of effective communication,
* Mentally healthy,
* Individuals who can comprehend and implement planned interventions before colonoscopy.

Exclusion Criteria:

* Individuals with a history of abdominal surgery,
* Those with serious illnesses that could affect the study outcomes (e.g., severe heart failure, kidney failure),
* Individuals using medications that could impact intestinal functions due to systemic diseases,
* Individuals who have not complied with the recommended interventions will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Classification (BBPS) | Day of colonoscopy only
  The Boston Bowel Preparation Scale (BBPS) is a rating scale used to evaluate the adequacy of bowel preparation.

SECONDARY OUTCOMES:
Patient satisfaction | 2 days
  The patient's perception of the usefulness of the intervention as self-reported in a preprocedural survey.

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim kiyat, Principal Investigator — PhD student
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data will be shared upon contact with researchers conducting meta-analysis or systematic reviews.